CLINICAL TRIAL: NCT03792776
Title: Effect of Lidocaine 1% and 2% in the Endotracheal Tube Cuff on Postoperative Sore Throat and Cough
Brief Title: Effect of Lidocaine 1% and 2% in the Tube Cuff on Postoperative Sore Throat and Cough
Acronym: ELIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ogarite Habib (Other)
Responsible Party: Sponsor-Investigator, Ogarite Habib, Principal Investigator, Saint-Joseph University
Organization: Saint-Joseph University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEHDF 1263
Record Dates: First submitted 2018-12-22; First posted 2019-01-03 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Sore Throat; Postoperative Cough
Keywords: Lidocaine 1%; Lidocaine 2%; Endotracheal tube cuff; Cuff inflation; Postoperative sore throat; Postoperative cough; General anesthesia; Endotracheal intubation
MeSH Terms: interventions — Air; Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Air (Active Comparator): Endotracheal tube cuff inflation with air
  Interventions: Other: cuff inflation with air; Other: Induction of anesthesia; Other: Maintenance of anesthesia; Other: Endotracheal intubation; Other: Systematic post-operative analgesia
- Lidocaine 1% (Experimental): Endotracheal tube cuff inflation with Lidocaine 1%
  Interventions: Drug: cuff inflation with lidocaine 1%; Other: Induction of anesthesia; Other: Maintenance of anesthesia; Other: Endotracheal intubation; Other: Systematic post-operative analgesia
- Lidocaine 2% (Experimental): Endotracheal tube cuff inflation with Lidocaine 2%
  Interventions: Drug: cuff inflation with lidocaine 2%; Other: Induction of anesthesia; Other: Maintenance of anesthesia; Other: Endotracheal intubation; Other: Systematic post-operative analgesia

INTERVENTIONS:
Other: cuff inflation with air — Endotracheal tube cuff inflation with air
  Arms: Air
Drug: cuff inflation with lidocaine 1% — Endotracheal tube cuff inflation with lidocaine 1%
  Arms: Lidocaine 1%
Drug: cuff inflation with lidocaine 2% — Endotracheal tube cuff inflation with lidocaine 2%
  Arms: Lidocaine 2%
Other: Induction of anesthesia — The induction of anesthesia will be made following a preoxygenation with a facial mask with 100% Oxygen. It consists on the intravenous injection of Sufentanil 5 mcg or Fentanyl 50mcg, Lidocaine 1mg/Kg, Propofol 2.5mg/kg, Rocuronium 0.6mg/kg or Cisatracurium 0.15mg/kg.
Other: Maintenance of anesthesia — Maintenance of anesthesia will be done by sevoflurane + nitrous oxide, and reinjections of morphinomimetics and curare will be made as needed (the total doses will be noted at the end of the intervention).
Other: Endotracheal intubation — The intubation is made by a N° 7.5 tube in men and a N° 7 tube in women. Cuff inflation will be done upon placement of the endotracheal tube. The cuff's pressure will be monitored at several intervals of the intervention and kept < or = 20 centimeter of water (cmH2O).
Other: Systematic post-operative analgesia — All patients will receive Paracetamol every 6 hours for the first 24 hours after the end of surgery.

SUMMARY:
Comparing the effect of different methods of endotracheal tube cuff inflation on the occurrence of a postoperative sore throat and cough (Air vs Lidocaine 1% vs Lidocaine 2%).

DETAILED DESCRIPTION:
Eligible patients undergoing general anesthesia will be randomized and assigned to three groups:

Group A: Endotracheal tube cuff inflation with air Group B: Endotracheal tube cuff inflation with Lidocaine 1% Group C: Endotracheal tube cuff inflation with Lidocaine 2%

The induction of anesthesia will be made following a preoxygenation with a facial mask with 100% Oxygen. It consists on the intravenous injection of Sufentanil 5 mcg or Fentanyl 50mcg, Lidocaine 1mg/Kg, Propofol 2.5mg/kg, Rocuronium 0.6mg/kg or Cisatracurium 0.15mg/kg.

Maintenance of anesthesia will be done by sevoflurane + nitrous oxide, and reinjections of morphinomimetics and curare will be made as needed (the total doses will be noted at the end of the intervention).

The intubation is made by a N° 7.5 tube in men and a N° 7 tube in women. Cuff inflation will be done upon placement of the endotracheal tube. The cuff's pressure will be monitored at several intervals of the intervention and kept < or = 20 centimeter of water (cmH2O).

The volume of lidocaine used will never exceed 5 mg / kg for the patient to be protected from the local toxicity of the local anesthetic in case of accidental rupture of the balloon.

All patients will receive Paracetamol every 6 hours for the first 24 hours after the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* American Society of Anesthesiologists classification (ASA) category 1 or 2
* High pressure, low volume endotracheal tube - (Lo-pro)

Exclusion Criteria:

* Ear nose and throat and cranial surgery
* Ear nose and throat pathologies
* Asthma and bronchial hyperreactivity
* Chronic cough
* Diabetes
* Cognitive disorders
* Swallowing disorders
* Corticotherapy during the last week
* Allergy to lidocaine
* Urgent surgery
* Nasogastric, oro-gastric
* Ventral position
* More than 2 intubation attempts
* Continuous intravenous infusion of lidocaine intraoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Sore throat intensity 0 | hour 0 after extubation
  Throat pain evaluation using the visual analog scale of pain (range from 0 cm (no pain) to 10 cm (very intense pain))
Sore throat intensity 2 | at 2 hours after extubation
  Throat pain evaluation using the visual analog scale of pain (range from 0 cm (no pain) to 10 cm (very intense pain))
Sore throat intensity 6 | at 6 hours after extubation
  Throat pain evaluation using the visual analog scale of pain (range from 0 cm (no pain) to 10 cm (very intense pain))
Sore throat intensity 24 | at 24 hours after extubation
  Throat pain evaluation using the visual analog scale of pain (range: from 0 cm (no pain) to 10 cm (very intense pain))
Cough intensity 0 | hour 0 after extubation
  Cough intensity evaluation using the visual analog scale of cough (range from 0 cm (no cough) to 10 cm (very severe cough))
Cough intensity 2 | at 2 hours after extubation
  Cough intensity evaluation using the visual analog scale of cough (range from 0 cm (no cough) to 10 cm (very severe cough))
Cough intensity 6 | at 6 hours after extubation
  Cough intensity evaluation using the visual analog scale of cough (range from 0 cm (no cough) to 10 cm (very severe cough))
Cough intensity 24 | at 24 hours after extubation
  Cough intensity evaluation using the visual analog scale of cough (range from 0 cm (no cough) to 10 cm (very severe cough))

CONTACTS AND LOCATIONS:
Overall Officials: Hicham Jabbour, MD, Study Director — Saint JU